CLINICAL TRIAL: NCT07076550
Title: A Phase 1-1b Study to Evaluate the Safety, Efficacy and Dosimetry of [225Ac]Ac-A9-3408 in Subjects With Unresectable or Metastatic Melanoma
Brief Title: A Phase 1-1b Study to Evaluate the Safety, Efficacy and Dosimetry of Study Drug A9-3408 in Subjects With Metastatic Melanoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Alpha-9 Oncology USA Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: A9-3408-01
Record Dates: First submitted 2025-06-27; First posted 2025-07-22 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Melanoma Metastatic; Uveal Melanoma, Metastatic; Mucosal Melanoma
Keywords: Metastatic Melanoma; Melanoma; Radiopharmaceuticals; Theranostic
MeSH Terms: conditions — Uveal Melanoma; Neoplasm Metastasis; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 Dose Escalation (Experimental): Participants enrolled in Dose Escalation will receive a single dose of the investigational diagnostic agent [68Ga]Ga-A9T-3202 during screening, and receive the investigational treatment [225Ac]Ac-A9-3408 once every 6 weeks, for up to 6 total cycles.
  Interventions: Drug: [225Ac]Ac-A9-3408; Diagnostic Test: [68Ga]Ga-A9T-3202
- Phase 1B Dose Expansion (Experimental): Participants enrolled in Dose Expansion will receive a single dose of the investigational diagnostic agent [68Ga]Ga-A9T-3202 during screening, and receive the investigational treatment [225Ac]Ac-A9-3408 once every 6 weeks, for up to 6 total cycles.
  Interventions: Drug: [225Ac]Ac-A9-3408; Diagnostic Test: [68Ga]Ga-A9T-3202

INTERVENTIONS:
Drug: [225Ac]Ac-A9-3408 — Administered IV
Diagnostic Test: [68Ga]Ga-A9T-3202 — Administered IV

SUMMARY:
The goal of this trial is to see if this investigational drug is safe for adult patients with melanoma that has spread to other parts of the body or cannot be removed by surgery. It will also see if this investigational drug can shrink melanoma tumors in the body. The main questions this study aims to answer are:

* What are the side effects of this investigational drug?
* What is the highest dose of this investigational drug that can be given safely?

Participants will:

* Take the investigational drug once every 6 weeks, for up to 6 times in total
* Visit a doctor's office on a regular basis for checkups and tests

DETAILED DESCRIPTION:
This is a multicenter, open-label Phase 1-1b study of [225Ac]Ac-A9-3408 in subjects with unresectable or metastatic melanoma.

The primary aim of the Phase 1 portion of the study is to evaluate the safety and tolerability as well as the normal organ and tumor dosimetry of [225Ac]Ac-A9-3408 and to select a recommended Phase 2 dose (RP2D).

The aim of Phase 1b will be to evaluate the safety, efficacy, and normal organ and tumor dosimetry of [225Ac]Ac-A9-3408 administered at the RP2D in subjects with unresectable or metastatic cutaneous melanoma who had confirmed disease progression while receiving an anti-PD-1/PD-L1-containing regimen.

The interventional diagnostic [68Ga]Ga-A9T-3202 will be administered intravenously (IV) once during screening.

The interventional drug [225Ac]Ac-A9-3408 will be administered intravenously (IV) once every 6 weeks, for a total of up to 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* [68Ga]Ga-A9T-3202 uptake in at least one measurable lesion (per RECIST v1.1) on PET scan
* Histologically or cytologically confirmed unresectable or metastatic melanoma with disease progression on prior standard of care therapy
* Adequate ECOG performance status
* Adequate baseline organ function within 14 days of first dose of investigational product
* Recovered from side effects of prior anticancer therapy
* Women of childbearing potential (WOCBP) must have a negative pregnancy test and follow adequate birth control method(s) during the treatment period and for at least 6 months after last dose of [225Ac]Ac-A9-3408. Sexually active males with partners who are WOCBP must agree to adequate birth control method(s) during the treatment period and for at least 3 months after last dose of [225Ac]Ac-A9-3408

Exclusion Criteria:

* Previous treatment with radioactive nuclides except radioactive imaging tracers
* Treatment with another investigational product shortly prior to first dose of [225Ac]Ac-A9-3408 with exception of anti-PD-1/PD-L1 agents.
* Concurrent anticancer therapy
* Major surgery within 4 weeks of first dose of investigational product
* Second malignancy within 2 years
* Active, clinically serious infection
* Known infusion reactions to components of the investigational product
* Other clinically serious health conditions including cardiovascular and or severe infectious diseases
* Significant central nervous system metastatic disease
* Pregnant, breastfeeding or unwilling to practice adequate birth control method(s)
* Any condition per the opinion of the investigator that would impact the safety of the subject, protocol adherence or ability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Determine max tolerated dose and recommended Phase 2 Dose | First 28 days following first study treatment
  Rate of DLTs per dose level/cohort
Incidence of treatment-related adverse events | From first study treatment until end of treatment
  Rate and severity of suspected treatment-related adverse events, change from baseline laboratory values and change from baseline vital signs as graded by CTCAE version 5.0

SECONDARY OUTCOMES:
Evaluate the preliminary efficacy of [225Ac]Ac-A9-3408 by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) | Up to 1 year from enrollment
  Percent of patients who achieve an overall response (ORR), defined as the percent of patients who achieve a complete response (CR) or partial response (PR) by RECIST v1.1
Evaluate biodistribution and normal organ dosimetry of [225Ac]Ac-A9-3408 | Up to 7 days following each cycle (42 days)
  Absorbed radiation dose estimates (Gy) in normal organs for [225Ac]Ac-A9-3408

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Alfred Health, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - GenesisCare Murdoch, Murdoch, Western Australia

IPD SHARING:
Plan to Share IPD: No